CLINICAL TRIAL: NCT00754325
Title: Phase II Randomized Trial of Fulvestrant With or Without Dasatinib in Men and Postmenopausal Women Who Have Hormone Receptor-positive Advanced Breast Cancer Previously Treated With an Aromatase Inhibitor
Brief Title: Randomized Trial of Fulvestrant With or Without Dasatinib in Men and Postmenopausal Women Who Have Hormone Receptor-positive Advanced Breast Cancer Previously Treated With an Aromatase Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-158; USOR 06-030
Record Dates: First submitted 2008-08-29; First posted 2008-09-17 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Dasatinib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Dasatinib +Fulvestrant) (Active Comparator)
  Interventions: Drug: Dasatinib; Drug: Fulvestrant
- Arm 2 (Fulvestrant) (Active Comparator)
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 100 mg, once daily (QD), upto 2 years
  Other Names: Sprycel
  Arms: Arm 1 (Dasatinib +Fulvestrant)
Drug: Fulvestrant — Intramuscular injection (IM), loading dose (500 mg) on Day 1 followed by 500 mg on Day 15 of Cycle 1. In subsequent cycles, 500 mg IM administered on Day 1. IM day 1 and 15 first cycle then IM Day 1 for all other cycles for 2 years
  Other Names: Faslodex

SUMMARY:
The purpose of this study is to find out what effect the combination of fulvestrant (Faslodex) and dasatinib (Sprycel) has on advanced breast cancer compared to fulvestrant alone.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb (BMS) clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Histologically confirmed hormone receptor positive (HR+) [(estrogen receptor (ER+) and/or progesterone receptors(PgR+)] breast cancer according to immunohistochemistry (IHC)
* Measureable or evaluable-only disease
* human epidermal growth factor receptor 2+ (HER2+) or HER2- breast cancer
* Males and females ≥18 years of age
* Females are post menopausal or surgically sterile
* Recurrent or progressive advanced breast cancer (locally-advanced or metastatic), that has progressed: (a) during or within 12 months after completion of adjuvant Aromatase Inhibitor (AI) treatment OR (b) during AI treatment in advanced setting (metastatic therapy)

Exclusion Criteria:

* Pregnant or breast feeding
* >1 chemotherapy regimen for advanced disease
* Pleural or pericardial effusion
* Serious cardiac condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-09; Primary Completion 2011-11 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (28):
- United States (28):
  - Northern Arizona Hematology & Oncology Associates, Sedona, Arizona
  - Arizona Oncol Assoc Dba (Hem Onc Physicians&Extenders) Hope, Tucson, Arizona
  - Florida Cancer Institute - New Hope, Hudson, Florida
  - Cancer Centers Of Florida, P.A, Ocoee, Florida
  - Central Indiana Cancer Centers, Carmel, Indiana
  - Kansas City Cancer Center, Llc., Overland Park, Kansas
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - New York Oncology Hematology, Pc, Troy, New York
  - Raleigh Hematology Oncology Associates, Raleigh, North Carolina
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Texas Oncology-Central Austin Cancer Center, Austin, Texas
  - Texas Oncology, P.A., Bedford, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Oncology, Dallas, Texas
  - Texas Oncology Sammons Cancer Center, Dallas, Texas
  - Texas Cancer Center, Denton, Texas
  - El Paso Cancer Treatment Ctr - West, El Paso, Texas
  - Us Oncology Research, Inc., Houston, Texas
  - Quest Diagnostic Clinical Laboratories Inc, Houston, Texas
  - Cancer Care Centers Of South Texas, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology Cancer Care And Research Center, Waco, Texas
  - Texas Oncology, P.A., Webster, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology & Hematology Associates Of Southwest Virginia, Inc., Salem, Virginia
  - Virginia Center Specialists, Pc, Woodbridge, Virginia

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started September 2008 and completed January 2014; 9 participants chose to remain on active treatment after the study completed.
Pre-assignment Details: 100 participants were enrolled and 100 participants were randomized (50 to each arm). 99 were treated (50 with fulvestrant + dasatinib and 49 with single-agent fulvestrant). Reason for non-treatment is that there was 1 withdrawal by participant.
Groups:
- Fulvestrant and Dasatinib: Arm 1: Participants in this group received a drug regimen that consisted of both fulvestrant and dasatinib.
  Fulvestrant: Intramuscular injection (IM), loading dose (500 mg) on Day 1 followed by 500 mg on Day 15 of Cycle 1 (28-day cycle). In subsequent cycles, 500 mg IM administered on Day 1, up to 2 years.
  Dasatinib: Tablets, Oral, 100 mg, once daily (QD), up to 2 years
- Fulvestrant: Arm 2: Participants in this group received a drug regimen that consisted of fulvestrant only.
  Fulvestrant: Intramuscular injection (IM), loading dose (500 mg) on Day 1 followed by 500 mg on Day 15 of Cycle 1 (28-day cycle). In subsequent cycles, 500 mg IM administered on Day 1, up to 2 years.
Period: Initial Treatment
Arm/Group | Fulvestrant and Dasatinib | Fulvestrant
Started | 50 | 49
Completed | 0 | 0
Not Completed | 50 | 49
Not completed — Continuing Active Treatment | 4 | 5
Not completed — Adverse Event | 7 | 6
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Sponsor Request | 0 | 1
Not completed — Disease Progression | 35 | 35
Period: Progression and Cross-over
Arm/Group | Fulvestrant and Dasatinib | Fulvestrant
Started | 0 (Arm 1 participants with dasatinib-related toxicity stop dasatinib, continue fulvestrant (Arm 1b).) | 21 (Progressive disease participants in Arm 2 could add dasatinib (Arm 2b) at investigator discretion.)
Completed | 0 | 0
Not Completed | 0 | 21

BASELINE CHARACTERISTICS:
Population: Intent To Treat (ITT) Population; all randomized participants
Groups:
- Fulvestrant and Dasatinib: Participants in this group received a drug regimen that consisted of both fulvestrant and dasatinib.
  Fulvestrant: Intramuscular injection (IM), loading dose (500 mg) on Day 1 followed by 500 mg on Day 15 of Cycle 1 (28-day cycle). In subsequent cycles, 500 mg IM administered on Day 1, up to 2 years.
  Dasatinib: Tablets, Oral, 100 mg, once daily (QD), up to 2 years
- Fulvestrant: Participants in this group received a drug regimen that consisted of fulvestrant only.
  Fulvestrant: Intramuscular injection (IM), loading dose (500 mg) on Day 1 followed by 500 mg on Day 15 of Cycle 1 (28-day cycle). In subsequent cycles, 500 mg IM administered on Day 1, up to 2 years.
- Total: Total of all reporting groups
Arm/Group | Fulvestrant and Dasatinib | Fulvestrant | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (12.3) | 61.4 (10.3) | 62.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 49 | 99
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Progression (PD) or Death
Description: This endpoint evaluated the progression free survival (PFS) of participants amongst the total evaluable population. Progression free survival (PFS) was defined as the time from randomization to either the date the subject was first recorded as having PD (even if the subject went off treatment because of toxicity), or the date of death if the subject died due to any causes before progression. Participants with no recorded post-baseline tumor assessment had PFS censored at the day of randomization. Participants lost to follow-up were censored at the last date of contact. Participants that had not progressed or died had PFS censored at the date of last follow-up.
Time Frame: Date of randomization to date of initial disease progression, or date of death (whichever occurs first), up to January 2014 (approximately 5 years)
Population: Evaluable population on initial treatment; all treated participants with measurable disease at baseline and at least one on-study tumor assessment. Participants without tumor response assessment due to rapid progression or study drug toxicity included as non-responders. Censored participants = 15 Fulvestrant and Dasatinib, 9 Fulvestrant
Measure: Number; unit: participants
Arm/Group | Fulvestrant and Dasatinib | Fulvestrant
Number analyzed (Participants) | 50 | 49
participants | 35 | 40

2. Secondary Outcome: Median Time of Progression-free Survival (PFS)
Description: Progression free survival (PFS) was defined as the time in months from randomization to either the date the subject was first recorded as having PD (even if the subject went off treatment because of toxicity), or the date of death if the subject died due to any causes before progression. Progression=At least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: as for outcome 1
Population: Evaluable population on initial treatment; all treated participants with measurable disease at baseline and at least one on-study tumor assessment. Participants without tumor response assessment due to rapid progression or study drug toxicity included in population as non-responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant and Dasatinib | Fulvestrant
Number analyzed (Participants) | 50 | 49
months | 5.6 [3.6 to 9.3] | 5.3 [3.0 to 7.4]

3. Secondary Outcome: Percentage of Participants With Progression Free Survival (PFS) at 6 Months
Description: PFS rate was defined as the percentage of participants experiencing no disease progression or death from any cause at 6 months after randomization. Progression free survival (PFS) was defined as the time from randomization to either the date the subject was first recorded as having PD (even if the subject went off treatment because of toxicity), or the date of death if the subject died due to any causes before progression. Progression=At least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Kaplan Meier assessments were used to estimate the percentages.
Time Frame: at 6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fulvestrant and Dasatinib | Fulvestrant
Number analyzed (Participants) | 50 | 49
percentage of participants | 48.1 [33.0 to 61.7] | 44.6 [30.1 to 58.1]

4. Secondary Outcome: Percentage of Participants With Clinical Benefit for At Least 6 Months
Description: Clinical benefit rate (CBR) was defined as the percentage of participants that had Stable Disease (SD), complete response (CR), or partial response (PR) for greater than or equal to 6 months if there was no evidence of progression at or before assessment performed on or after Study Day 161. CR= Disappearance of all target lesions. No new lesions. PR= At least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. SD= Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) taking as reference the smallest sum LD since the treatment started. Physical examination, radiological assessment, and bone scans (if applicable) were used to assess outcome.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fulvestrant and Dasatinib | Fulvestrant
Number analyzed (Participants) | 50 | 49
percentage of participants | 38.0 [24.7 to 52.8] | 42.9 [28.8 to 57.8]

5. Secondary Outcome: Number of Participants With Complete Response (CR) , Partial Response (PR), Stable Disease (SD), and Disease Progression (PD)
Description: Table represents the best response achieved over this time frame. CR = Disappearance of all target lesions. No new lesions. PR = At least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. SD = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) taking as reference the smallest sum LD since the treatment started. Progression (PD): At least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Fulvestrant and Dasatinib | Fulvestrant
Number analyzed (Participants) | 50 | 49
participants
  Complete Response, CR | 0 | 0
  Partial Response, PR | 1 | 3
  Stable Disease, SD | 34 | 28
  Disease Progression, PD | 11 | 16
  Not Evaluable | 4 | 2

6. Secondary Outcome: Number of Participants With Best Overall Response
Description: Best overall response rate (ORR) = number of participants with measurable lesions by Response Evaluation Criteria in Solid Tumors (RECIST) having a best response of complete response (CR) or partial response (PR) divided by number of randomized participants. RECIST 1.1 response criteria applies. To be recorded as best response, CR or PR had to be confirmed at ≥ 4 weeks interval. An unconfirmed CR was recorded as PR.
Time Frame: as for outcome 1
Population: Evaluable population on initial treatment with measurable lesion by RECIST (Response Evaluation Criteria In Solid Tumors). Participants without tumor response assessment due to rapid progression or study drug toxicity included in population as non-responders.
Measure: Number; unit: participants
Arm/Group | Fulvestrant and Dasatinib | Fulvestrant
Number analyzed (Participants) | 31 | 37
participants | 1 | 2

7. Secondary Outcome: Number of Participants With Serious Adverse Events, Death, and Discontinuation Due to Adverse Events
Description: Adverse event (AE) defined: any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Serious adverse event (SAE) defined: a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: as for outcome 1
Population: Safety Population on initial treatment; any participants that was randomized to any treatment group in the study and received at least one treatment therapy.
Measure: Number; unit: participants
Arm/Group | Fulvestrant and Dasatinib | Fulvestrant
Number analyzed (Participants) | 50 | 49
participants
  Serious Adverse Events | 14 | 11
  Deaths | 15 | 16
  Discontinued due to AEs | 7 | 6

ADVERSE EVENTS:
Time Frame: Date of randomization to date of initial disease progression, or date of death (whichever occurs first), up to January 2014 (approximately 5 years)
Description: Study initiated: September 2008; Study Completion: January 2014
Groups:
- Fulvestrant Crossover to Fulvestrant and Dasatinib: Arm 2b: Participants in this group started on the Fulvestrant only arm and later started receiving a drug regimen that consisted of both fulvestrant and dasatinib. These participants are all inclusive and not limited to Fulvestrant or Fulvestrant and Dasatinib treatment only. The timeframe for when these events occurred were not immediately available and may have been caused by previous exposure to Fulvestrant only (pre-crossover), therefore the events for this patient population are also reported separately.
  Fulvestrant: Intramuscular injection (IM), loading dose (500 mg) on Day 1 followed by 500 mg on Day 15 of Cycle 1 (28-day cycle). In subsequent cycles, 500 mg IM administered on Day 1, up to 2 years.
  Dasatinib: Tablets, Oral, 100 mg, once daily (QD), up to 2 years
Arm/Group | Fulvestrant and Dasatinib | Fulvestrant | Fulvestrant Crossover to Fulvestrant and Dasatinib
Serious Adverse Events (participants affected / at risk) | 14/50 | 11/49 | 7/21
Other Adverse Events (participants affected / at risk) | 48/50 | 44/49 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant and Dasatinib (N=50) | Fulvestrant (N=49) | Fulvestrant Crossover to Fulvestrant and Dasatinib (N=21)
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0
Hypertension (Cardiac disorders) | 1 | 0 | 0
Coagulation Time Increased (Cardiac disorders) | 0 | 1 | 0
Weakness Generalized (General disorders) | 0 | 1 | 1
Bowel Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Nausea and Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Obstruction Bowel (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Pancreatitis (Hepatobiliary disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Fracture Bone (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fracture Pathological (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Blackout Spell (Nervous system disorders) | 0 | 1 | 1
Brain metastases (Nervous system disorders) | 1 | 0 | 0
CSF Abnormal (Nervous system disorders) | 1 | 0 | 0
Chest Pain (Nervous system disorders) | 1 | 1 | 1
Chest Pain Substernal (Nervous system disorders) | 1 | 0 | 0
Pain (Nervous system disorders) | 1 | 0 | 0
Cough Productive (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Effusion Pleural (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Embolus Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pneumonia Lobar (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Stenosis Bronchial (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0
Urinary Tract Infection (Renal and urinary disorders) | 0 | 1 | 0
Thrombosis Venous Deep (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant and Dasatinib (N=50) | Fulvestrant (N=49) | Fulvestrant Crossover to Fulvestrant and Dasatinib (N=21)
Anemia (Blood and lymphatic system disorders) | 13 | 7 | 5
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 7 | 2 | 1
Effusion Pericardial (Cardiac disorders) | 3 | 0 | 0
Fatigue (General disorders) | 20 | 15 | 10
Weakness Generalized (General disorders) | 4 | 0 | 0
Weight Loss (General disorders) | 4 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 6 | 6
Hot Flashes (Endocrine disorders) | 4 | 6 | 1
Anorexia (Gastrointestinal disorders) | 6 | 6 | 4
Constipation (Gastrointestinal disorders) | 10 | 9 | 5
Diarrhea (Gastrointestinal disorders) | 19 | 8 | 7
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 2
Gastroesophageal Reflux (Gastrointestinal disorders) | 3 | 2 | 1
Nausea (Gastrointestinal disorders) | 23 | 12 | 8
Vomiting (Gastrointestinal disorders) | 8 | 7 | 6
Fever (Infections and infestations) | 5 | 4 | 2
Infection (Infections and infestations) | 3 | 0 | 0
Edema (Immune system disorders) | 4 | 2 | 1
Swelling (Immune system disorders) | 3 | 0 | 0
AST Increased (Metabolism and nutrition disorders) | 3 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 5 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 6 | 3
Joint Pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Pain Bone (Musculoskeletal and connective tissue disorders) | 5 | 4 | 2
Anxiety (Nervous system disorders) | 4 | 3 | 2
Depression (Nervous system disorders) | 4 | 4 | 1
Dizziness (Nervous system disorders) | 1 | 3 | 2
Headache (Nervous system disorders) | 10 | 8 | 5
Insomnia (Nervous system disorders) | 4 | 5 | 4
Chest Pain (Nervous system disorders) | 4 | 2 | 2
Injection Site Pain (Nervous system disorders) | 0 | 3 | 1
Pain (Nervous system disorders) | 17 | 16 | 11
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 11 | 2 | 1
Common Cold (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Coughing (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 5
Effusion Pleural (Respiratory, thoracic and mediastinal disorders) | 16 | 7 | 7
Infection Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.